CLINICAL TRIAL: NCT01155141
Title: Idiopathic Focal Segmental Glomerulosclerosis (FSGS) and Treatment With ACTH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-08182009-3600
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases

ARMS (1):
- No arms (Experimental): There are no arms to this study. All patients receive drug (H.P. Acthar Gel)
  Interventions: Drug: H.P. Acthar Gel

INTERVENTIONS:
Drug: H.P. Acthar Gel — Patients were treated with 40 units subcutaneously (SC) weekly for 2 weeks, then dose increased to 80 units SC weekly for 2 weeks followed by 80 units SC twice weekly to complete 16 weeks of therapy.

SUMMARY:
FSGS is an immunologic disorder wherein circulating immune proteins cause damage to the kidneys and progressive injury and scarring. Corticosteroid therapy is occasionally, but not nearly universally, successful in reducing proteinuria, and when patients respond, they have a favorable prognosis. The investigators believe that ACTH therapy (H.P. Acthar Gel) can provide a more rapid, well tolerated reduction in glomerular injury.

DETAILED DESCRIPTION:
EXPERIMENTAL TREATMENT: Patients with biopsy proven FSGS will be treated with ACTH in an open-label pilot study of tolerability and efficacy. The investigators will recruit 18-20 patients to complete this study, over 2 years.

ACTH therapy: Patients will receive H.P. Acthar gel IM or SQ, initially at 40 IU SQ every week for 16 weeks of therapy. All patients will be treated to goal BP of <140/90mmHg with all patients treated with ACEi or ARB therapy as tolerated. H2 receptor blockade or proton pump inhibitor therapy will also be offered all patients. Dose will be titrated up to 160 IU SQ every week, if at 1 month the patient has had no substantial reduction in proteinuria, no deterioration of blood pressure and no development of hyperglycemia as well as no serious adverse events felt to be related to the medication.

CLINICAL OUTCOME: Patients will be followed for the primary outcome of remission of proteinuria. This will be defined as partial remission when the proteinuria is reduced below 50% of the initial, pre treatment value and as complete remission when the proteinuria is reduced to < 0.5 g/g or <500 mg/day on a 24 hour urine sample. Secondary outcomes will include effects on eGFR, effects on glucose levels, effects on blood pressure (total doses of antihypertensive medications and absolute changes in blood pressure) and on immune status. Outcomes will be determined by looking at 3 month and 6 month values of urine protein and eGFR following initiation of treatment.

IMMUNOLOGIC TESTING: In order to further assess the role of immunologic perturations on FSGS and the effect of ACTH on the immune system, all patients will bank blood and urine before the start of the study for cytokine analysis, RNA, DNA, protein and protoarray testing.

MONITORING AND SAFETY: All patients will undergo full informed consent per the Stanford Institutional Review Board. Contact numbers will be provided and study staff will be available at all times in case of any medical emergencies. All patients will continue with routine health monitoring with a minimal of monthly assessments. A comprehensive interview will be undertaken to assess for side effects, complete physical exams will be accomplished including vital signs, CBC, clinical chemistries (including electrolytes, creatinine, glucose and liver function tests), urine for protein and creatinine and fasting lipid profiles every 3 months. Also at screening and baseline.

PATIENT WITHDRAWAL/TERMINATION OF STUDY: Patients will be closely monitored, as detailed above. Patients may voluntarily leave the study at any time, although every effort will be made to follow their clinical course and monitor for safety issues and possible benefits of therapy. Patient will be monitored for adverse events. Patients with severe adverse events will be evaluated for the relatedness of their event to the study medication. If the event is considered severe and possibly or probably related to the study medication, the medication will be discontinued and the patient will continue to be monitored. In the case the adverse event is possibly related, the medication may be restarted, if the investigator and subject agree. For patients with probably related severe adverse events, study treatment will be discontinued however, the investigators will still follow the patient to see if the course of their underlying disease was modified by treatment. As this is an open label, pilot study, no data safety monitoring board is felt to be necessary. If drug related SAEs develop in more than 20% of patients, the study will be submitted back to the IRB to determine if it should continue.

ELIGIBILITY:
Inclusion Criteria:

* 1. Biopsy proven FSGS
* 2. Ability to consent and complete study evaluations
* 3. Greater than 2g/day of proteinuria
* 4. No contraindications to treatment with corticosteroids or ACTH
* 5. Women of childbearing potential will agree to use effective forms of birth control throughout this study

Exclusion Criteria:

* 1. Known secondary cause of FSGS
* 2. Receiving active immune therapy (within 90 days)
* 3. Pregnancy
* 4. Creatinine >2.5 mg/dl
* 5. Uncontrolled HTN (>180/100mm Hg)
* 6. Diabetes
* 7. Acute or chronic infection
* 8. Severe comorbidity (active coronary, cerebrovascular disease, cancer, psychiatric disease)
* 9. Age < 16, >65 years
* 10. Evidence of untreated tuberculosis (+PPD or Ellispot Gold testing)
* 11. A known contraindication to ACTH. Corticotropin is considered contraindicated in patients with scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history of or the presence of a peptic ulcer, congestive heart failure, uncontrolled hypertension, or sensitivity to proteins of porcine origin.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lafayette, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Hogan J, Bomback AS, Mehta K, Canetta PA, Rao MK, Appel GB, Radhakrishnan J, Lafayette RA. Treatment of idiopathic FSGS with adrenocorticotropic hormone gel. Clin J Am Soc Nephrol. 2013 Dec;8(12):2072-81. doi: 10.2215/CJN.02840313. Epub 2013 Sep 5. PMID 24009220

RESULTS

PARTICIPANT FLOW:
Groups:
- H.P. Acthar Gel: Patients treated with 40 units subcutaneously (SC) weekly for 2 weeks, 80 units SC weekly for 2 weeks, then 80 units SC twice weekly to complete 16 weeks of therapy.
Period: Overall Study
Arm/Group | H.P. Acthar Gel
Started | 16
Completed | 14
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | H.P. Acthar Gel
Number analyzed (Participants) | 15
Age, Continuous [Median (Standard Deviation); unit: years] | 40 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
24 hour proteinuria [Median (Standard Deviation); unit: g/day] | 3.6 (5.7)
Serum Creatinine [Median (Standard Deviation); unit: mg/dL] | 1.4 (0.9)
Protein/creatinine ratio [Median (Standard Deviation); unit: unitless] | 3.1 (2.3)
Glucose [Median (Standard Deviation); unit: mg/dL] | 95 (8.4)
Weight [Median (Standard Deviation); unit: kg] | 87.3 (24.3)
Systolic blood pressure [Median (Standard Deviation); unit: mm Hg] | 128 (15.9)
Diastolic blood pressure [Median (Standard Deviation); unit: mm Hg] | 82 (9.8)
Total cholesterol [Median (Standard Deviation); unit: mg/dL] | 236 (99.5)
eGFR [Median (Standard Deviation); unit: mL/min/1.73m^2] | 56 (34.8)

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Proteinuria
Time Frame: Baseline - Month 6
Measure: Median (Standard Deviation); unit: g/day
Arm/Group | H.P. Acthar Gel
Number analyzed (Participants) | 15
g/day
  Baseline (N=15) | 3.6 (5.7)
  Week 5 (N=15) | 3.8 (8.6)
  Week 16 (N=14) | 2.2 (4.7)
  Month 6 (N=12) | 3.0 (3.2)

2. Primary Outcome: Serum Creatinine
Time Frame: Baseline - Month 6
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | H.P. Acthar Gel
Number analyzed (Participants) | 15
mg/dL
  Baseline (N=15) | 1.4 (0.9)
  Week 5 (N=15) | 1.8 (0.8)
  Week 9 (N=14) | 1.8 (1)
  Week 16 (N=14) | 1.9 (0.9)
  Month 6 (N=12) | 2.0 (1.1)

3. Secondary Outcome: eGFR
Time Frame: Baseline - Month 6
Measure: Median (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | H.P. Acthar Gel
Number analyzed (Participants) | 15
mL/min/1.73m^2
  Baseline (N=15) | 56.0 (34.8)
  Week 5 (N=15) | 44.0 (37.1)
  Week 9 (N=14) | 37.5 (32.0)
  Week 16 (N=14) | 43.0 (28.0)
  Month 6 (n=12) | 38.0 (33.5)

4. Primary Outcome: Protein/Creatinine Ratio
Time Frame: Baseline - Month 6
Measure: Median (Standard Deviation); unit: unitless
Arm/Group | H.P. Acthar Gel
Number analyzed (Participants) | 15
unitless
  Baseline (N=15) | 3.1 (2.3)
  Week 5 (N=15) | 3.1 (5.3)
  Week 16 (N=14) | 2.4 (1.8)
  Month 6 (N=11) | 1.6 (1.3)

5. Secondary Outcome: Weight
Time Frame: Baseline - Month 6
Measure: Median (Standard Deviation); unit: kg
Arm/Group | H.P. Acthar Gel
Number analyzed (Participants) | 15
kg
  Baseline (N=15) | 87.5 (24.3)
  Week 5 (N=15) | 89.8 (24.7)
  Week 9 (N=13) | 94.0 (25.2)
  Week 16 (N=13) | 93.8 (26.1)
  Month 6 (N=11) | 91.3 (28.2)

6. Secondary Outcome: Systolic Blood Pressure
Time Frame: Baseline - Month 6
Measure: Median (Standard Deviation); unit: mm Hg
Arm/Group | H.P. Acthar Gel
Number analyzed (Participants) | 15
mm Hg
  Baseline (N=15) | 128.0 (15.9)
  Week 5 (N=15) | 136.0 (15.2)
  Week 9 (N=13) | 136.0 (18.3)
  Week 16 (N=14) | 134.0 (18.6)
  Month 6 (N=11) | 128.0 (15.6)

7. Secondary Outcome: Diastolic Blood Pressure
Time Frame: Baseline - Month 6
Measure: Median (Standard Deviation); unit: mm Hg
Arm/Group | H.P. Acthar Gel
Number analyzed (Participants) | 15
mm Hg
  Baseline (N=15) | 82.0 (9.8)
  Week 5 (N=15) | 85.0 (11.1)
  Week 9 (N=13) | 80.0 (10.1)
  Week 16 (N=14) | 78.0 (12.1)
  Month 6 (N=11) | 77.0 (8.4)

8. Secondary Outcome: Glucose
Time Frame: Baseline - Month 6
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | H.P. Acthar Gel
Number analyzed (Participants) | 15
mg/dL
  Baseline (N=15) | 95 (8.4)
  Week 5 (N=15) | 92.0 (14.9)
  Week 9 (N=14) | 93.0 (24.0)
  Week 16 (N=14) | 97.0 (17.2)
  Month 6 (N=13) | 88.0 (14.3)

9. Secondary Outcome: Total Cholesterol
Time Frame: Baseline - Month 6
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | H.P. Acthar Gel
Number analyzed (Participants) | 14
mg/dL
  Baseline (N=15) | 236.0 (99.5)
  Week 5 (N=14) | 215.0 (86.2)
  Week 16 (N=13) | 229.0 (90.4)
  Month 6 (N=13) | 217.0 (133.3)

ADVERSE EVENTS:
Arm/Group | H.P. Acthar Gel
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | H.P. Acthar Gel (N=15)
Hyperglycemia (Metabolism and nutrition disorders) | 1 — grade 3
Acute Kidney Injury (Renal and urinary disorders) | 1 — grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | H.P. Acthar Gel (N=15)
Elevated Blood Pressure (Vascular disorders) | 2 — Grade 1
Altered Mood (Psychiatric disorders) | 1 — Grade 1
Increased Energy (Metabolism and nutrition disorders) | 4 — Grade 1
Vertigo (Ear and labyrinth disorders) | 1 — Grade 1
Slow Wound Healing (Skin and subcutaneous tissue disorders) | 1 — Grade 1
Bruising at Injection Site (Injury, poisoning and procedural complications) | 1 — Grade 1
Nausea (Gastrointestinal disorders) | 1 — Grade 1
Increased Appetite (Metabolism and nutrition disorders) | 1 — Grade 1
Cold (Infections and infestations) | 1 — Grade 1
Fatigue (General disorders) | 2 — Grade 1
Weight Gain (Investigations) | 2 — One patient had grade 1 weight gain, another patient had grade 2 weight gain
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 1 — Grade 1
Headache (Nervous system disorders) | 1 — Grade 1
Polyuria (Renal and urinary disorders) | 1 — Grade 1
Rash (Skin and subcutaneous tissue disorders) | 1 — Grade 1
Facial Swelling (General disorders) | 1 — Grade 2
Leg Swelling (General disorders) | 2 — Grade 1
Acne (Skin and subcutaneous tissue disorders) | 3 — 2 patients had grade 1 acne, one patient had grade 2 acne.
Cushingoid (Endocrine disorders) | 1 — grade 1
Nephrotic Syndrome (Renal and urinary disorders) | 1 — grade 2
Felt Faint after Injection (Nervous system disorders) | 1 — grade 1
Hypokalemia (Metabolism and nutrition disorders) | 1 — grade 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 — grade 1
Blurred Vision (Eye disorders) | 1 — grade 1
Right Arm Numbness (Nervous system disorders) | 1 — grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No